CLINICAL TRIAL: NCT06934785
Title: The Combination of Letrozole (LE) and Clomiphene Citrate (CC) or LE Alone for Ovulation Induction in Women With WHO Group II/IV Ovulatory Disorders: A Randomized Controlled Trial
Brief Title: LE + CC vs. LE for Ovulation Induction
Acronym: COLA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mỹ Đức Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02/25/DD/BVMD
Record Dates: First submitted 2025-04-07; First posted 2025-04-18 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Letrozole; Clomiphene Citrate; Ovulation Disorder; Ovulation Induction
MeSH Terms: interventions — Sex

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination of LE and CC group (Active Comparator): 5 milligrams LE per day (Femara® 2.5 milligrams, Novartis, Switzerland) and 50 milligrams CC (Duinum 50 milligrams, Medochemie, Cyprus) per day, starting on the second to the fourth day of the cycle, for five consecutive days.
  Interventions: Procedure: IUI or intercourse
- LE alone group (Active Comparator): 5 milligrams LE per day (Femara® 2.5 milligrams, Novartis, Switzerland), starting on the second to the fourth day of cycle, for five consecutive days.
  Interventions: Procedure: IUI or intercourse

INTERVENTIONS:
Procedure: IUI or intercourse — 5 milligrams LE per day (Femara® 2.5 milligrams, Novartis, Switzerland) and 50 milligrams CC (Duinum 50 milligrams, Medochemie, Cyprus) or 5 milligrams LE per day (Femara® 2.5 milligrams, Novartis, Switzerland) will be started on the second to the fourth day of the cycle, for five consecutive days. An ultrasound will be carried out three days after the last dose of medicine (day 8 of OI) to evaluate ovarian follicles' growth and the endometrium's thickness. If the follicular diameter reach ≥14 millimetres, check-up will be planned every two days until it reaches 18 millimetres. If there is the appearance of at least one follicle reaching 18 millimetres or more, a human chorionic gonadotropin (hCG) injection (IVF-C 5000 IU, LG Life Science, Korea) will be administered on the same day of the ultrasound in order to induce ovulation. IUI will be scheduled 36 - 38 hours after hCG injection or intercourse will be scheduled in the next day.

SUMMARY:
This randomized controlled trial (RCT) aims to evaluate whether, in infertile women with WHO II/IV ovulatory disorders, a combination of letrozole (LE) and clomiphene citrate (CC) compared to LE alone, result in higher live birth rates.

The study is designed as an open-label, multicenter RCT across six fertility clinics in Vietnam. Participants will be randomized into two groups: (1) LE + CC , (2) LE alone. The primary outcome measure is the live birth rate after one treatment cycle. Based on prior data, the live birth rate for IUI in letrozole cycles is estimated at 12%. To detect a 10% increase in live birth rates with CC, 436 couples are needed (α = 0.05, power = 80%). Additionally, the live birth rate after IUI with LE-induced ovulation is approximately 18.7% (Diamond et al., 2015). To detect a 10% increase with CC, 560 couples are required (α = 0.05, power = 80%). Considering a 5% loss to follow-up and protocol deviations, the study plans to recruit 600 participants (150 per arm).

DETAILED DESCRIPTION:
Letrozole (LE) has been suggested as a first-line treatment for ovulation induction in PCOS. Clomiphene citrate (CC) is another widely used drug to induce ovulation in women with PCOS. Due to the different mechanisms of action of CC and letrozole, it is possible that taking these drugs together may increase the ovulation rate by having a synergistic effect with their own mechanisms and resulting to increase the pregnancy outcome of patients undergoing ovulation induction (OI).

Mejia et al. conducted a randomized controlled trial (RCT) and reported the ovulation rate was significantly higher in the combination group than in the LE-alone group (N=70, 77% vs. 42.9%, respectively; RR 1.80 95%. CI. 1.18 to 2.75, P=0.007). This finding is confirmed by another RCT but not in a third more recent RCT, with larger sample size. Live birth rate was only reported as secondary endpoint in two studies, with a non-significant difference between the two groups [12% vs. 7%, RR 1.68, 95% CI 0.19 to 14.66) and 16.4% vs. 18.6%, RR 0.92, 95% CI 0.57 to 1.50)]. Therefore, we plan an RCT to evaluate whether a combination of LE and CC results in higher live birth rates than LE alone in women with WHO II/IV ovulatory disorders.

This is a open-label, multicenter, randomized controlled trial across six fertility clinics in Vietnam. Potentially eligible participants will be given a study information sheet during their first consultation, at least 2 weeks before the start of the menstrual cycle, whether spontaneous or induced. In case the women present to the clinic during their menstrual cycle and wish to start treatment straightaway, they will be given the information sheet to read while waiting for the clinicians. Screening for eligibility will be performed by treating physicians on the day OI starts. Eligible participants will be invited to a full discussion with investigators about the study. Women who fulfil the eligibility criteria and who have been counselled before will be formally invited to participate in the study. If the women agree to participate, they will be asked to sign the informed consent form. After informed consent, a fasting blood sample will be obtained for hormone and biochemical analysis.

Participants will be randomized in a 1:1 ratio to receive the combination of LE and CC (LE+CC) and LE alone. The computer-generated random list will be prepared by an independent statistician who has no other involvement in the study. Assignment to treatment allocation will be done via a web portal hosted by HOPE Research Center, Vietnam. The randomization schedule will be computer-generated at HOPE Research Center, with a permuted random block size of 4 and 8.

Combination of LE and CC group: 5 milligrams LE per day (Femara® 2.5 milligrams, Novartis, Switzerland) and 50 milligrams CC (Duinum 50 milligrams, Medochemie, Cyprus) per day, starting on the second to the fourth day of the cycle, for five consecutive days.

LE alone group: 5 milligrams LE per day (Femara® 2.5 milligrams, Novartis, Switzerland), starting on the second to the fourth day of cycle, for five consecutive days.

IUI or natural intercourse will be indicated based on the physicians and patients.

The primary endpoint will be live birth after one treatment cycle.

ELIGIBILITY:
Inclusion Criteria:

* Women 18-40 years of age
* Having WHO II/IV ovulatory disorders (length of cycle < 21 or > 35 days or having < 8 cycles per year)
* Progressive motility (PR) ≥ 32%, sperm concentration ≥ 5 million/ml, total progressive motility sperm count > 5 million (World Health Organization, 2021)
* Written informed consent.
* Not participating in other studies.

Exclusion Criteria:

* Untreated thyroid disease; Thyroid disease is suspected if patients have one of these (Bednarczuk et al., 2021); TSH ≥4 mIU/L or TSH ≥2.5mIU/L and TPOAb (+) or TSH <0.1mIU/L
* Untreated hyper-prolactinemia; Hyperprolactinemia is suspected if patients have prolactinemia concentration >50 ng/mL (The sample is collected after an overnight fast, at least 2 hours after waking up, ensuring that venipuncture does not cause excessive stress.)
* Allergy or having contraindications to LE or CC;
* Unilateral or Bilateral fallopian tube blockage (HSG, HyFoSy or surgery confirmation)
* Untreated endometrial abnormalities include endometrial hyperplasia, intrauterine adhesions, endometrial polyp, or chronic endometritis.
* Uterine abnormalities include leiomyomas L0, L1, or L2; severe adenomyosis; congenital uterine abnormalities, include didelphus, arcuate, unicornuate, bicornuate, septate.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Live birth after one treatment cycle | At 22 weeks of gestation
  Live birth will be defined as the complete expulsion or extraction from a woman of a product of fertilization, after 22 completed weeks of gestational age; which, after such separation, breathes or shows any other evidence of life, such as heart beat, umbilical cord pulsation or definite movement of voluntary muscles, irrespective of whether the umbilical cord has been cut or the placenta is attached.

SECONDARY OUTCOMES:
Duration of stimulation | During the intervention
  Duration of stimulation
Number of follicles ≥14mm on day of hCG | During the intervention
  Number of follicles ≥14mm on day of hCG
Endometrial thickness on day of hCG | During the intervention
  Endometrial thickness on day of hCG
Cycle cancellation | At 21 day of the ovulation induction cycle
  The cycle will be cancelled if (1) there is no follicle reaches ≥18 millimetres) on day 21 of the OI; (2) there are ≥ 3 follicles with diameter ≥16 millimetres or (3) ≥ 4 ovarian follicles with diameter ≥10 millimetres
Ovulation | At day 7 after the hCG injection
  A serum midluteal progesterone (17-OH-progesterone) will be measured on day 7 after the hCG injection. A level of >3 ng/mL (>9.5 nmol/L) will be used as evidence of ovulation.
Positive pregnancy test | At day 15 after IUI or timed intercourse
  Serum human chorionic gonadotropin level greater than 25 mIU/mL at day 15 after IUI or timed intercourse
Clinical pregnancy | After 6 weeks of gestation
  Diagnosed by ultrasonographic visualization of one or more gestational sacs or definitive clinical signs of pregnancy at 6 weeks or more. In addition to intra-uterine pregnancy, it includes a clinically documented ectopic pregnancy
Ongoing pregnancy | After 12 weeks of gestation
  Pregnancy with a detectable heart rate at 12 weeks gestation or beyond
Multiple pregnancies | At 6-9 weeks of gestation
  The presence of more than one sac at early pregnancy ultrasound (6-9 weeks gestation)
Multiple birth | At 22 weeks of gestation
  The complete expulsion or extraction from a woman of more than one fetus, after 22 completed weeks of gestational age, irrespective of whether it is a live birth or stillbirth
Ectopic pregnancy | At 7 weeks of gestation
  A pregnancy outside the uterine cavity, diagnosed by ultrasound, surgical visualization or histopathology
Miscarriage <22 weeks | Before 22 completed weeks of gestation
  Spontaneous loss of pregnancy up to 22 weeks of gestation
Gestational age at delivery | At the time of delivery
  Gestational age at delivery
Growth restriction | At the time of delivery
  a birth weight < 10th percentile
Stillbirth | After 20 completed weeks of gestational age
  The death of a fetus prior to the complete expulsion or extraction from its mother after 20 completed weeks of gestational age. The death is determined by the fact that, after such separation, the fetus does not breathe or show any other.
Premature birth | At 22, 28, 32 weeks and 37 weeks of gestation
  Multiple definitions, defined as delivery at <24, <28, <32, <37 completed weeks
Onset of labour | At the time of delivery
  Onset of labour
Mode of delivery | At the time of delivery
  Mode of delivery
Birth weight | At the time of delivery
  Weight of singletons and twins
Low birth weight | At the time of delivery
  Weight < 2500 gm at birth
Very low birth weight | At the time of delivery
  Weight < 1500 gm at birth
High birth weight | At the time of delivery
  Weight 4000 gm or 4500 gm at birth
Very high birth weight | At the time of delivery
  Weight over than 4.500 g for women with diabetes, and a threshold of 5000 g for women without diabetes
Gestational diabetes mellitus | At 24 to 28 weeks of gestation
  GDM is diagnosed using a 75g oral glucose tolerance test
Hypertension in pregnancy | after 20 weeks of gestation or beyond
  Pregnancy-induced hypertension, pre-eclampsia, eclampsia and HELLP syndrome
Congenital abnormalities | At birth
  Structural or functional disorders that occur during intra-uterine life and can be identified prenatally, at birth or later in life. Congenital anomalies can be caused by single gene defects, chromosomal disorders, multifactorial inheritance, environmental teratogens, and micronutrient deficiencies. The time of identification should be reported
Neonatal mortality | within 28 days of birth
  Death of a live-born baby within 28 days of birth
NICU admission | At birth
  The admittance of the newborn to NICU
Reported side-effects | During the intervention
  included headache, hot flashes, abdominal bloating, abdominal pain including cramps, nausea, mood changes, fatigue, back pain, dizziness, breast discomfort, diarrhoea, night sweats, sleep disturbances
Hospitalized or seek any additional care during the ovulation induction cycle | During the intervention
  Hospitalized or seek any additional care during the ovulation induction cycle
Incidence of Ovarian hyperstimulation syndrome (OHSS) | 10 days after the intervention
  A potentially lethal iatrogenic complication of the early luteal phase or/and early pregnancy after OI or ovarian stimulation. OHSS was evaluated if symptoms were reported by the patient. OHSS was classified using the flow diagram

CONTACTS AND LOCATIONS:
Overall Officials: Lan N Vuong, PhD,MD, Principal Investigator — University of Medicine and Pharmacy at Ho Chi Minh City
Locations (1):
- My Duc Hospital, Ho Chi Minh City, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Teede HJ, Tay CT, Laven JJE, Dokras A, Moran LJ, Piltonen TT, Costello MF, Boivin J, Redman LM, Boyle JA, Norman RJ, Mousa A, Joham AE. Recommendations From the 2023 International Evidence-based Guideline for the Assessment and Management of Polycystic Ovary Syndrome. J Clin Endocrinol Metab. 2023 Sep 18;108(10):2447-2469. doi: 10.1210/clinem/dgad463. PMID 37580314
- [Background] Weiss NS, Nahuis MJ, Bordewijk E, Oosterhuis JE, Smeenk JM, Hoek A, Broekmans FJ, Fleischer K, de Bruin JP, Kaaijk EM, Laven JS, Hendriks DJ, Gerards MH, van Rooij IA, Bourdrez P, Gianotten J, Koks C, Lambalk CB, Hompes PG, van der Veen F, Mol BWJ, van Wely M. Gonadotrophins versus clomifene citrate with or without intrauterine insemination in women with normogonadotropic anovulation and clomifene failure (M-OVIN): a randomised, two-by-two factorial trial. Lancet. 2018 Feb 24;391(10122):758-765. doi: 10.1016/S0140-6736(17)33308-1. Epub 2017 Dec 19. PMID 29273245
- [Background] Mejia RB, Summers KM, Kresowik JD, Van Voorhis BJ. A randomized controlled trial of combination letrozole and clomiphene citrate or letrozole alone for ovulation induction in women with polycystic ovary syndrome. Fertil Steril. 2019 Mar;111(3):571-578.e1. doi: 10.1016/j.fertnstert.2018.11.030. Epub 2019 Jan 22. PMID 30683591
- [Background] Diamond MP, Legro RS, Coutifaris C, Alvero R, Robinson RD, Casson P, Christman GM, Ager J, Huang H, Hansen KR, Baker V, Usadi R, Seungdamrong A, Bates GW, Rosen RM, Haisenleder D, Krawetz SA, Barnhart K, Trussell JC, Ohl D, Jin Y, Santoro N, Eisenberg E, Zhang H; NICHD Reproductive Medicine Network. Letrozole, Gonadotropin, or Clomiphene for Unexplained Infertility. N Engl J Med. 2015 Sep 24;373(13):1230-40. doi: 10.1056/NEJMoa1414827. PMID 26398071